CLINICAL TRIAL: NCT06448000
Title: Impact of Storage Time in Liquid Nitrogen on Cryopreserved Human Spermatozoa
Brief Title: Effect of Long-time Human Sperm Storage in Liquid Nitrogen on Semen Parameters
Acronym: CRYOFERT
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 20220911-CRYOFERT
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-03

CONDITIONS: Healthy; Cancer; Infertility, Male; Cryopreservation
Keywords: Cryopreservation; semen standard parameters; liquid nitrogen; high security straws; long term storage; progressive and total mobility
MeSH Terms: conditions — Neoplasms; Infertility, Male

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Same semen samples are analyzed in group 1 and 2. Group 1 correspond to ejaculate semen samples analyzed the day of slow-freezing
- Group 2: Same semen samples are analyzed in group 1 and 2. Group 2 correspond to the same ejaculate semen samples as group 1 but analyzed after a storage time from 2 to 12 years in liquid nitrogen.

SUMMARY:
Sperm cryopreservation is an essential tool for men fertility preservation in the context of gonadotoxic treatments or/and pathologies such as cancers, gamete donation and ART. Nevertheless, it is validated that the freezing and thawing procedures affect sperm parameters and in particular motility. It is therefore essential to determine the impact of storage time on motility and particularly the number of progressive motile spermatozoa which will determine the choice of ART technique. However, few studies have analyzed the impact of storage time in liquid nitrogen and no study over a long period on human spermatozoa and their use in ART.

The aim of this study is to assess the impact of long-time storage, from 2 to 12 years, in liquid nitrogen on standard semen parameters, notably motility.

DETAILED DESCRIPTION:
It has been demonstrated in the literature that cryopreservation of semen samples in liquid nitrogen guaranty good post thawing motility recovery. However, the literature is scarce and relatively old. Moreover, studies only described very small samples cohort and do not specify in which container the samples are stored. There are currently no published studies on high security straws which are widely used for semen cryopreservation worldwide.

The aim of this study is to assess the impact of long-time storage, from 2 to 12 years, in high security straws, in liquid nitrogen on human standard semen parameters, notably on motility.

Hundred and one cryopreserved semen samples between 2010 to 2020 were donated to research by patients monitored in the unit of Assisted Reproductive Technology - Conservation of human sperm and eggs (ART-CECOS) Unit of the University Hospital of Clermont-Ferrand for fertility preservation. Only samples corresponding to the inclusion criteria below were included in the study without distinction of bio clinical criteria.

All analyzed samples have been cryopreserved following the same protocol, in high security 0,3ml straws, with the same cryoprotectant and using the same programmable freezer Nanodigitcool (CryoBiosystem).

The day of cryopreservation, a post-freezing test (T0) was caried by thawing a straw and by assessing sperm count, motility and vitality according to WHO guidelines 2010.

After a storage time from 2 to 12 years, a second post-freezing test (T1) was caried by thawing two straws and by assessing sperm count, motility and vitality in the same way as T0.

The statistical difference, concordance, correlation and diagnostic agreement between T0 and T1 were analyzed.

This study is the first to assess the integrity of human sperm after a long-time cryopreservation in liquid nitrogen on a large cohort (more than 100 samples).

ELIGIBILITY:
Inclusion Criteria:

* The ejaculates were frozen in high security straws by slow freezing,
* At least two straws per sample were available
* The "post-freezing" thawing test was carried out on the day of freezing
* The "post-freezing" thawing test carried out at T0 includes cell numbering, vitality and mobility
* There is the informed signature of the consent to donate the straws to Research by the patient

Exclusion Criteria:

* Ejaculate not donated to research, lack of consent to donation to research
* Frozen ejaculate in microdrop
* Thawing test not carried out or incomplete

Ages: 19 Years to 63 Years | Sex: Male
Age Groups: Adult
Study Population: All samples frozen between 2010 and 2020 corresponding to the inclusion criteria cited above have been included in the study.
  In total, this corresponds to 101 eligible samples, or 202 straws, between 2010 and 2020, i.e. a T1 storage time studied from 2 to 12 years.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
To evaluate and compare the total and progressive mobility of human spermatozoa post-freezing and post-storage in High Security straws. | 07/2022 to 03/2023
  The percentage of total and progressive motile human spermatozoa were assessed according to WHO, 2010 guideline.

SECONDARY OUTCOMES:
To compare the vitality of post-freezing and post-storage human spermatozoa | 07/2022 to 03/2023
  The percentage of alive human spermatozoa were assessed according to WHO, 2010 guideline.
To compare the number of motile, total and progressive spermatozoa post-freezing and post-storage | 07/2022 to 03/2023
  The number of motile human spermatozoa were assessed according to WHO, 2010 guideline.

CONTACTS AND LOCATIONS:
Overall Officials: Hanae Pons-Rejraji, PhD, Principal Investigator — University Hospital, Clermont-Ferrand; Florence Brugnon, MD, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- University Hospital, Clermont-Ferrand, France